CLINICAL TRIAL: NCT05094869
Title: Prevention of HCC Using Mobile Phone Applications: A Disease Management Project Based on CR-HepB Platform
Brief Title: Prevention of HCC Using Mobile Phone Applications
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jidong Jia, Director of Liver Research Center, Beijing Friendship Hospital
Other Study IDs: YYYXYJ-2021-182
Record Dates: First submitted 2021-09-22; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Liver Cirrhosis; Hepatitis B
Keywords: Compensatory hepatitis B cirrhosis; Health management; Mobile health application; Compliance
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- APP self-management group: Patients would register on the APP and visit the clinics according to the routine practice and guidelines. During the study, the APP would regularly send messages including the follow-up reminder (manually set up by the patients on the APP), medication reminder, health education knowledge, etc.
  Interventions: Behavioral: Use of mobile health application; Behavioral: Self follow-up reminders
- APP intelligent-management group: Patients would register on the APP and visit the clinics according to the routine practice and guidelines. During the study, the APP would regularly send messages including the follow-up reminder (automatically set up by the APP), medication reminder, health education knowledge, etc. The doctors will evaluate their disease progression every six months through the APP and guide patients' clinical practice accordingly.
  Interventions: Behavioral: Use of mobile health application; Behavioral: Online interaction; Behavioral: Intelligent follow-up reminders
- Control group: History data of another 4000 Patients who have been on the platform of China Registry of Hepatitis B (CR-Hep B) and been diagnosed as compensatory hepatitis B cirrhosis would be extracted and serve as the control group (No APP, no follow-up reminders, no online interaction).

INTERVENTIONS:
Behavioral: Use of mobile health application — The APP would regularly send messages including the medication reminder, health education knowledge, etc.
  Groups: APP intelligent-management group; APP self-management group
Behavioral: Online interaction — The patients would be able to upload their examination results in the APP and then the doctors will evaluate their disease progression every six months through the APP and guide patients' clinical practice accordingly.
  Groups: APP intelligent-management group
Behavioral: Self follow-up reminders — The APP would regularly send messages including the follow-up reminder (manually set up by the patient on the APP)
  Groups: APP self-management group
Behavioral: Intelligent follow-up reminders — The APP would regularly send messages including the follow-up reminder (automatically set up by the APP)
  Groups: APP intelligent-management group

SUMMARY:
This prospective cohort study is initiated to evaluate the compliance improvement to the standardized follow-up and clinical management in the population of compensatory hepatitis B cirrhosis with a mobile health application (APP). Patients were enrolled and divided into APP self-management group (APP only ) and APP intelligent-management group (APP and online interaction). The compliance to the standardized follow-up and clinical management (every six months) under the two clinical management modes would be evaluated and compared with the history data extracted from the platform of China Registry of Hepatitis B (CR-Hep B).

DETAILED DESCRIPTION:
Standardized follow-up and clinical management in the population of compensatory hepatitis B cirrhosis is important in the prevention of liver cancer. In the clinical practice, follow-up every six months are usually recommended. This prospective cohort study is initiated to evaluate the compliance improvement to the standardized follow-up and clinical management with a health management application (APP). 4000 patients who have registered on the platform of China Registry of Hepatitis B (CR-Hep B) and been diagnosed as compensatory hepatitis B cirrhosis would be recruited in the study. They were divided into two groups according to whether they use the APP and whether there is online interaction between doctors and patients:

1. APP self-management group (APP only, N=1000): Patients would register on the APP and visit the clinics according to the routine practice and guidelines. During the study, the APP would regularly send messages including the follow-up reminder (manually set up by the patients on the APP), medication reminder, health education knowledge, etc.
2. APP intelligent-management group (APP and online interaction, N=3000): Patients would register on the APP and visit the clinics according to the routine practice and guidelines. During the study, the APP would regularly send messages including the follow-up reminder (automatically set up by the APP), medication reminder, health education knowledge, etc. The doctors will evaluate their disease progression every six months through the APP and guide patients' clinical practice accordingly.

Patients in these two groups would be followed up for 2 years after enrollment. Besides, history data of another 4000 Patients who have been on the platform of China Registry of Hepatitis B (CR-Hep B) and been diagnosed as compensatory hepatitis B cirrhosis would be extracted and serve as the control group (No APP and No online interaction, N=4000).

The compliance to the standardized follow-up and clinical management (every six months) under the three clinical management modes would be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Registered on the CR-HepB platform
* Requiring or receiving antiviral therapy using nucleoside (acid) analogues (recommended as the first-line therapy in the 2019 Chinese Guidelines for Chronic Hepatitis B Prevention and Treatment )
* Diagnosed as compensatory hepatitis B cirrhosis, with the diagnostic criteria fitting any of the following criteria:

  1. Diagnosis of Liver cirrhosis by histology;
  2. Varicose veins in Esophageal and/or gastric fundus indicated by endoscopy;
  3. Diagnosis of Liver cirrhosis by Imaging examination (abdominal ultrasound, CT, MRI) ;
  4. Liver elasticity measurement >12.0 kpa (ALT<5×ULN)
  5. Platelet PLT lower than the lower limit of normal value, and Serum albumin (ALB) lower than 35 g/L or international standardized ratio (INR) >1.3.
* Completing the informed consent form

Exclusion Criteria:

* With any decompensated cirrhosis events, such as esophagogastric variceal rupture and bleeding, ascites, and hepatic encephalopathy;
* With any malignant tumor;
* With serious illness on any vital organs and systems, including heart, lungs, kidneys, and blood;
* Unsuitable for participating the study deemed by researchers;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 4000 patients who have registered on the platform of China Registry of Hepatitis B (CR-Hep B) and been diagnosed as compensatory hepatitis B cirrhosis would be recruited in the study. Besides, history data of another 4000 Patients who have been on the platform of China Registry of Hepatitis B (CR-Hep B) and been diagnosed as compensatory hepatitis B cirrhosis would be extracted and serve as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient compliance to the standardized semi-annual follow-up | 0 to 2 years
  Total follow-up times with the three clinical management modes. The event of follow-up is defined as self-reported clinic visit for liver cirrhosis assessment on the mobile phone application by patients.

SECONDARY OUTCOMES:
Applicability of mobile phone application | 0 to 2 years
  Applicability of mobile phone application is defined as cumulative minutes of APP use over the study period, which is recorded by APP itself.
Clinical performance on HCC of the three clinical management modes | 0 to 2 years
  Clinical performance on HCC is defined as the proportion of early stage HCC among all detected HCC. The event of HCC is measured with self-reported HCC and the stage on the mobile phone application by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jidong Jia, MD, PhD, Principal Investigator — Beijing Friendship Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] Yang B, Zhang B, Xu Y, Wang W, Shen Y, Zhang A, Xu Z. Prospective study of early detection for primary liver cancer. J Cancer Res Clin Oncol. 1997;123(6):357-60. doi: 10.1007/BF01438313. PMID 9222303
- [Background] Singal AG, Pillai A, Tiro J. Early detection, curative treatment, and survival rates for hepatocellular carcinoma surveillance in patients with cirrhosis: a meta-analysis. PLoS Med. 2014 Apr 1;11(4):e1001624. doi: 10.1371/journal.pmed.1001624. eCollection 2014 Apr. PMID 24691105
- [Background] Marrero JA, Kulik LM, Sirlin CB, Zhu AX, Finn RS, Abecassis MM, Roberts LR, Heimbach JK. Diagnosis, Staging, and Management of Hepatocellular Carcinoma: 2018 Practice Guidance by the American Association for the Study of Liver Diseases. Hepatology. 2018 Aug;68(2):723-750. doi: 10.1002/hep.29913. No abstract available. PMID 29624699
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of alcohol-related liver disease. J Hepatol. 2018 Jul;69(1):154-181. doi: 10.1016/j.jhep.2018.03.018. Epub 2018 Apr 5. No abstract available. PMID 29628280